CLINICAL TRIAL: NCT06037330
Title: Analgesic Effect and Safety Analysis of Nalbuphine in ARDS Patients After Surgery
Brief Title: Nalbuphine in ARDS Patients After Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hairong Chen (Other)
Responsible Party: Sponsor-Investigator, Hairong Chen, Doctor of Medicine（M.D.）, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QFSYXLL-KY-2022(092)
Record Dates: First submitted 2023-08-17; First posted 2023-09-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Nalbuphine; Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nalbuphine group (Experimental): 40 mg of nalbuphine was diluted into 50 mL solution, the load dose was 0.1mg/kg, the maintenance dose was 0.04-0.08mg/kg/h, the CPOT score was <2, and the daily maximum dose was 160mg.
  Interventions: Drug: Nalbuphine
- Sufentanil group (Active Comparator): 0.1mg of sufentanil was diluted into 50 mL solution, the loading dose was 0.2-0.5μg/kg, the maintenance dose was 0.2-0.3μg/kg/h, and the CPOT score was <2 points.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Nalbuphine — Nalbuphine was injected intravenously. The target CPOT score was <2, and the target RASS score was -2 ~ 1. 40 mg of nalbuphine was diluted into 50 mL solution, the load was 0.1mg/kg, the maintenance dose was 0.04-0.08mg/kg/h, the CPOT score was <2, and the maximum daily dose was 160mg.
  Other Names: Nalbuphine Hydrochloride Injection
  Arms: Nalbuphine group
Drug: Sufentanil — Sufentanil was injected intravenously, and the target CPOT score was <2, and the target RASS score was -2 ~ 1. 0.1mg of sufentanil was diluted into 50 mL solution, the loading dose was 0.2-0.5μg/kg, the maintenance dose was 0.2-0.3μg/kg/h, and the CPOT score was <2 points
  Other Names: Sufentanil citrate Injection
  Arms: Sufentanil group

SUMMARY:
Critically ill patients need reasonable and moderate analgesic and sedative treatment to eliminate or reduce pain, anxiety and restlessness, improve patient comfort and cooperation, reduce patients' stress response, protect organ function and optimize prognosis. As a semi-synthetic opioid receptor agonist-antagonist, nalbuphine can bind to μ, κand δ receptors, has partial antagonistic effect on μ receptor, and is fully activated on κreceptor, with very weak δ receptor activity. Results of a study on the efficacy and safety of nalbuphine for analgesia in ICU patients showed that nalbuphine has sustained and stable analgesic effect for patients with mild to moderate analgesic needs in ICU, the onset time is comparable to sufentanil, and excessive sedation caused by sufentanil can be avoided, and the effect on hemodynamics is small. It can be used as a new choice of analgesic drugs in ICU.

A single-center, randomized, single-blind, prospective study was designed to compare nalbuphine and sufentanil in patients with ARDS after surgery. Sixty patients with ARDS after surgery to be admitted to ICU were randomly divided into experimental group (Nalbuphine group) and control group (Sufentanil group). This study aims to determine the analgesic efficacy and safety of nalbuphine hydrochloride in patients with Acute Respiratory distress syndrome (ARDS) after surgery. The successful development of this study will provide more theoretical basis for the individualized analgesic sedation program for surgical patients.

DETAILED DESCRIPTION:
Severe patients need reasonable and moderate analgesic sedation to eliminate or reduce pain, anxiety and agitation, improve comfort and cooperation, reduce stress response, protect organ function and improve prognosis. As a semi-synthetic opioid receptor agonist-antagonist, nalbuphine can bind to μ, κand δ receptors, has partial antagonistic effect on μ receptor, and is fully activated on κreceptor, with very weak δ receptor activity. Nalbuphine exerts powerful analgesic and sedative effects at the spinal cord level, with rapid analgesic effect and long duration, almost no cardiovascular adverse reactions, mild respiratory depression and capping effect, low incidence of nausea, vomiting and skin pruritus, and low addiction. Results of a study on the efficacy and safety of nalbuphine for analgesia in ICU patients showed that nalbuphine has sustained and stable analgesic effect for patients with mild to moderate analgesic needs in ICU, the onset time is comparable to sufentanil, and excessive sedation caused by sufentanil can be avoided, and the effect on hemodynamics is small. It can be used as a new choice of analgesic drugs in ICU. Moreover, nalbuphine theoretically has no σ-receptor excitability, is not hallucinogenic, and the chance of inducing delirium is lower. Studies have shown that nalbuphine can reduce postoperative inflammation and oxidative stress and has a lung protective effect.

This study aims to determine the analgesic efficacy and safety of nalbuphine hydrochloride in patients with Acute Respiratory distress syndrome (ARDS) after surgery, and to explore the effects of nalbuphine hydrochloride on respiratory function, gastrointestinal function and cognitive function. To provide more theoretical basis for individualized analgesic and sedation program for surgical patients. Sixty patients were included and randomly divided into 1:1 groups, with 30 patients in each group. All patients were included according to strict inclusion criteria.

The experimental group was given nalbuphine analgesia and the control group was given sufentanil analgesia. The number of patients reaching the target level of analgesia and sedation at each time node, invasive mechanical ventilation time, oxygenation index change, mortality and other indicators were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Had undergone surgical treatment within 7 days before enrollment;
* Meet the diagnostic criteria for ARDS proposed at the 2011 Berlin ARDS Definition Conference;
* Age ≥18 years old, gender unlimited;
* Patients admitted to ICU with CPOT score ≥3;
* Stay in ICU ≥48h;
* Sign the informed consent form.

Exclusion Criteria:

* APACHE II score ≥23 points;
* Patients with esophageal reflux disease and severe gastrointestinal injury have AGI score ≥3;
* Long-term use of narcotic analgesics, hypnotics and psychotropic drugs;
* Alcohol withdrawal symptoms;
* Severe liver dysfunction (Child-Pugh grade C);
* Patients with bronchial asthma and myasthenia gravis;
* Patients with severe craniocerebral injury, brain tumor, and increased intracranial pressure are prone to respiratory depression;
* Patients undergoing cardiac surgery under cardiopulmonary bypass;
* Patients who have been enrolled in other clinical trials;
* Study patients with drug allergy or other contraindications;
* Pregnant or lactating women;
* The patient himself or his legally authorized representative is unwilling to sign the informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number 1 of patients who achieved the target level of analgesia and sedation | 30 minutes after the analgesic is administered
  The number of patients in the two groups who reached the target level of analgesia and sedation within 30 minutes after the administration of analgesic drugs was compared
Number 2 of patients who achieved the target level of analgesia and sedation | 60 minutes after the analgesic is administered
  The number of patients in the two groups who reached the target level of analgesia and sedation within 60 minutes after the administration of analgesic drugs was compared
Number 3 of patients who achieved the target level of analgesia and sedation | 4 hours after the analgesic is administered
  The number of patients in the two groups who reached the target level of analgesia and sedation within 4 hours after the administration of analgesic drugs was compared
Number 4 of patients who achieved the target level of analgesia and sedation | 8 hours after the analgesic is administered
  The number of patients in the two groups who reached the target level of analgesia and sedation within 8 hours after the administration of analgesic drugs was compared
Number 5 of patients who achieved the target level of analgesia and sedation | 12 hours after the analgesic is administered
  The number of patients in the two groups who reached the target level of analgesia and sedation within 12 hours after the administration of analgesic drugs was compared
Number 6 of patients who achieved the target level of analgesia and sedation | 24 hours after the analgesic is administered
  The number of patients in the two groups who reached the target level of analgesia and sedation within 24 hours after the administration of analgesic drugs was compared
Comparison of invasive mechanical ventilation time | The time from the start of the tracheal intubation to the withdrawal of the ventilator, assessed up to 28 days
  Invasive mechanical ventilation time was compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Hairong Chen, doctor, Study Director — Qianfo Mountain Hospital, Shandong Province
Locations (1):
- Department of Intensive Care Medicine, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zacny JP, Conley K, Galinkin J. Comparing the subjective, psychomotor and physiological effects of intravenous buprenorphine and morphine in healthy volunteers. J Pharmacol Exp Ther. 1997 Sep;282(3):1187-97. PMID 9316825